CLINICAL TRIAL: NCT05008822
Title: Effect of Motor Imaginary Training on Upper Limb Functions in Stroke Patients
Brief Title: Effect of Motor Imaginary Training on Upper Limb Functions in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/0832 Zulfiqar Ali
Record Dates: First submitted 2021-08-03; First posted 2021-08-17 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Stroke, Cardiovascular
Keywords: Motor imaginary technique
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imaginary Training Group (Experimental): After the baseline assessment, the participant will receive Motor Imaginary Program
  Interventions: Other: Motor Imaginary Training Group
- Task oriented Training Group (Active Comparator): After the baseline assessment, the participant will receive MRP and CIMT training
  Interventions: Other: Task oriented Training Group

INTERVENTIONS:
Other: Motor Imaginary Training Group — After the baseline assessment, the participant will receive Motor Imaginary Program
  Arms: Motor Imaginary Training Group
Other: Task oriented Training Group — After the baseline assessment, the participant will receive MRP and CIMT training
  Arms: Task oriented Training Group

SUMMARY:
This study will provide knowledge about effectiveness of motor imaginary training in upper limb performance in chronic stroke patients. Very little data is available about the use in Motor Imaginary in post stroke upper limb rehabilitation in Pakistan. Moreover, studies done previously did not specified population of stroke; This study will include MCA stroke patients only, whom upper limb weakness is more prevalent.

DETAILED DESCRIPTION:
Motor imagery is a technique for inducing motor activity in response to a certain motor output by producing a mental image of the action without intending to conduct it. It is a cognitive technique that, rather than making a patient to pick up new procedures, promotes neural alterations in order enable the patient to re-acquire motor skills mastered before the CVA or copy the actions of others. Motor imaging training is a sort of therapy in which the patient imagines a gesture or movement in order to learn, reinforce, or improve the movement's performance. A study done in South Korea, published in 2015, revealed that Motor imagery training has a good impact on UL performance by refining functional mobility during stroke rehabilitation. The results suggest that motor imagery training is viable and helpful for improving UL function in CVA patients.

Meta-analysis done in Australia in the year 2013, was supportive of Motor imaginary techniques further convincing that Mental imagery can be a possible intervention for stroke patients given that it being, safe cost-effective & unlimited practice opportunities. Study done in China in 2017, suggested that clinicians should consider the use of MI in addition to treatment currently used to improve upper extremity functions after stroke as no evidence of side effects or harm was noted . RCT done in year 2006 in USA indicated that for patients with chronic, moderate upper limb impairment after CVA, program of CIMT with mental practice only resulted in decrease impairment, with functional enhancement.

ELIGIBILITY:
Inclusion Criteria:

* MCA stroke
* Chronic stroke patients
* Mini-Mental State Examination (MMSE) score >24 points
* Spasticity grade II and III on Modified Ashworth scale

Exclusion Criteria:

* Severe cognitive disability such as depression, unilateral neglect, seizure, dementia,
* Any MSK disorder including muscle contracture

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
wolf motor function | Change from Baseline to 4th Weeks
  The Wolf Motor Function Test (WMFT) is a timed and functional test that assesses upper extremity motor skills in a quantitative manner.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah ghous, MS, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Physical therapy department of Rehman Medical Institute, Peshawar, Pakistan, Peshawar, Khyber Pakhtunkha, Pakistan

IPD SHARING:
Plan to Share IPD: No